CLINICAL TRIAL: NCT03777254
Title: A Double-center, Open-label,Single Ascending Dose Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Intravitreous Injections of RC28-E (a Chimeric Decoy Receptor Trap Fusion Protein by Dual Blockage of VEGF and FGF-2) in Subjects With Wet Age-Related Macular Degeneration
Brief Title: Evaluation the Pharmacokinetics,Safety,Tolerability of Single Intravitreal Injection RC28-E in Subjects With Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C001AMDCLLI
Record Dates: First submitted 2018-12-09; First posted 2018-12-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — RC28-E protein; Fibroblast Growth Factor 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RC28-E (Experimental): "·Experimental:RC28-E 0.25mg Injection:single Intravitreal Injection Intervention: Biological: RC28-E
  * Experimental: RC28-E 0.5mg Injection:single Intravitreal Injection Intervention: Biological: RC28-E
  * Experimental: RC28-E 1.0mg Injection:single Intravitreal Injection Intervention: Biological: RC28-E
  * Experimental: RC28-E 2.0mg Injection:single Intravitreal Injection Intervention: Biological: RC28-E"
  Interventions: Biological: RC28-E

INTERVENTIONS:
Biological: RC28-E — RC28-E intravitreous injection 50ul
  Other Names: RC28-E is a chimeric decoy receptor trap fusion protein by dual blockage of VEGF and FGF-2.

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety, tolerability and pharmacokinetics of single intravitreous injections,single ascending doses, of RC28-E(a chimeric decoy receptor trap fusion protein by dual blockage of VEGF and FGF-2) in subjects with wet age-related macular degeneration (wAMD).

DETAILED DESCRIPTION:
This is an open-label, non-randomized,double-center phase 1 study evaluating pharmacokinetics, safety and tolerability of single intravitreal injections of RC28-E in the patients with AMD.RC28-E is recombinant dual decoy receptor IgG1 Fc-fusion protein,can block VEGF-A and FGF-2. In preclinical studies suggested that RC28-E might be more effective in inhibiting pathological angiogenesis than other VEGF antagonists on CNV. Every subject will only accept one dose. In addition to safety and preliminary efficacy, pharmacokinetics and immunogenicity of RC28-E will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal representative signed informed consent;
2. Aged 50 years to 80 years, male or female;
3. Best corrected VA for the studied eye≥34 letters, ≤73 letters(By ETDRS chart);
4. With choroidal neovascular (CNV) lesions secondary to neovascular AMD;
5. If both eyes meet the criteria, severe illness eye will be selected; if both eyes are the same, the right eye will be selected as the study eye.

Exclusion Criteria:

1. History of any vitreous hemorrhage with 2 months prior to screening;
2. Presence of scar, fibrosis or atrophy in central foveal of the study eye;
3. Significant refractive media opacity, including cataract, may interfere with visual assessment;
4. The studied eye suffered pseudoexfoliation syndrome, central retinal vein occlusion, intraocular hemorrhage resulting in decreased vision, rhegmatogenous retinal detachment, macular hole, choroidal neovascularization (CNV) for any reason other than AMD (such as fundus angioid streaks, ocular histoplasmosis, pathologic myopia, trauma);
5. Afferent pupillary defect(APD);
6. The intraocular pressure is higher than 25mmHg despite medication treatment;
7. Active infectious conjunctivitis, keratitis, scleritis, uveitis and endophthalmitis;
8. Best corrected VA for the studied eye≤19 letters(By ETDRS chart);
9. Topical or grid photocoagulation within 3 months before screening;
10. Uncontrolled diabetes mellitus(fast glucose level≥7.0 mmol/L or ≥11.1 mmol/L 2h after meal;
11. The studied eye received any intraocular surgery or laser treatment (such as macular translocation surgery, glaucoma filtering surgery, transpupillary thermotherapy, foveal photocoagulation surgery, vitrectomy, optic neurotomy, optic nerve sheath fenestration; But cataract surgery, verteporfin photodynamic therapy, Nd:YAG laser posterior capsulotomy more than 3 months before screening can be selected;
12. Any eye or whole body received anti-angiogenic drug such as pegaptanib, Aflibercept, Ranibizumab, Bevacizumab,conbercept within 3 months before baseline visit;
13. Any eye received intraocular injection of corticosteroid drugs (such as triamcinolone acetonide) within 3 months before screening, or periocular injection of corticosteroid drugs within 1 months before screening;
14. Allergic to sodium fluorescein, indocyanine green, therapeutic or diagnostic protein products, and allergic ≥2 drugs and/or non-drugs, or with current allergic diseases;
15. With surgery within one month prior to enrollment, or with unhealed wound, ulcer, fracture at present;
16. No lens (excluding intraocular lens);
17. Uncontrolled hypertension(defined as those who received the best treatment regimen, >180 mmHg systolic was measured once, >160 mmHg systolic or > 100 mmHg diastolic was measured twice in succession);
18. With a history of myocardial infarction within 6 months before screening;
19. With activity disseminated intravascular coagulation and significant bleeding tendency prior to screening; Using anticoagulants or antiplatelet aggregation drugs in addition to aspirin/NSAIDs within 14 days before screening;
20. Any uncontrolled clinical disease (such as severe mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant tumors);
21. Pregnant (blood pregnancy test positive) and lactating women and patients who cannot take effective contraception(such as intrauterine devices, acyeterion, condoms, etc.) between study period or 30 days after visit;
22. Patients who participated in or were currently attending other clinical studies within 30 days before screening;
23. The patients is considered unsuitable for enrollment by investigator. "

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular and systemic adverse events and serious adverse events which are related to RC28-E | 42 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve(AUC) | 42 days
Maximum observed maximum plasma concentration (Cmax) | 42 days
Time to reach the maximum observed plasma concentration (Tmax) | 42 days
T1/2(Terminal phase half life after single dose) | 42 days
Change in Best Corrected Visual Acuity (BCVA) from baseline | 42 days
Change in Central Retinal Thickness（CRT）from baseline | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: wenbin wei, Principal Investigator — BEIJING TONGREN HOSPITAL.CMU
Locations (1):
- Beijing Tongren Hospital .Cmu, Beijing, China

REFERENCES:
- [Derived] Kou X, Sun Y, Li S, Bian W, Liu Z, Zhang D, Jiang J. Pharmacology Study of the Multiple Angiogenesis Inhibitor RC28-E on Anti-Fibrosis in a Chemically Induced Lung Injury Model. Biomolecules. 2019 Oct 24;9(11):644. doi: 10.3390/biom9110644. PMID 31652997